CLINICAL TRIAL: NCT03864250
Title: Tacrolimus Monotherapy for Idiopathic Membranous Nephropathy: A Randomized, Open, Controlled, Multicenter Clinical Trial
Brief Title: Tacrolimus Monotherapy for Idiopathic Membranous Nephropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XH-19-002
Record Dates: First submitted 2019-03-04; First posted 2019-03-06 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-03

CONDITIONS: Tacrolimus; Idiopathic Membranous Nephropathy; Clinical Trial
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — Tacrolimus; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tacrolimus monotherapy (Experimental)
  Interventions: Drug: Tacrolimus
- Tacrolimus combined with hormone therapy (Active Comparator)
  Interventions: Drug: Tacrolimus; Drug: Prednisone

INTERVENTIONS:
Drug: Tacrolimus — The initial dose of TAC is 0.05-0.1 mg/kg/d, taking 2 hours before and after meals. The interval is strictly 12 hours. The blood concentration is measured after taking the drug. According to the concentration of blood drug valley, the dose of tacrolimus (blood concentration of ≤10ng/ml) is adjusted. If the blood drug concentration is low, the drug dose (≤0.1mg/kg/d) is increased accordingly. After 6 months of treatment, the drug is discontinued. The TAC dose is maintained at the original dose after 6 months of treatment with complete or partial remission of urinary protein until the end of the 48-week trial.
Drug: Prednisone — The initial dose of prednisone is 0.5 mg/kg/d orally (maximum dose 40 mg/d), and after 8-12 weeks, the dose was gradually reduced until discontinuation. TAC treatment is given at the same time (the treatment plan is the same as the experimental group).
  Arms: Tacrolimus combined with hormone therapy

SUMMARY:
This random, open, control and multicenter clinical trial mainly aims to assess the urine protein remission rate of tacrolimus (TAC) monotherapy for idiopathic membranous nephropathy (IMN).

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 - 80 years;
2. Those whose clinical manifestation and renal biopsy pathologic diagnosis are IMN (Stages I-IV) with secondary membranous nephropathy excluded;
3. Those who meet any of the following high-risk IMN standards:

   * Urinary protein>8g/24h
   * Serum albumin<25g/l
   * Serum PLA2R levels are 5 times higher than normal
   * eGFR decline rate after confirmed IMN within 6-12 months is ≥30%
   * Patients with serious complications: pulmonary embolism, lower extremity static Vein thrombosis/embolism, acute renal injury, etc.
4. Those without reaching the above high-risk IMN standard, but their course of disease is >6 months without spontaneous remission,and still present nephrotic syndrome;
5. Patients who have signed the informed consent forms.

Exclusion Criteria:

1. Those whose kidney pathological manifestation of interstitial fibrosis is >30%;
2. Those who are positive in active Hepatitis B (including HBsAg, HBeAg and HBcAb or HBsAg, HBeAb and HBC) or serological indexes (HBsAg or/and HBeAg or/and HBcAb) or infected with Hepatitis C, tuberculosis, cytomegalovirus, severe fungal infection, syphilis or HIV infection;
3. Those who suffer from untreated active digestive tract ulcer within 3 months before random grouping;
4. Those who suffer from uncured malignant tumor less than 5 years;
5. Those who received glucocorticoids (prednisone or prednisolone), mycophenolate mofetil, tacrolimus, cyclosporine A, cyclophosphamide, tripterygium and other immunosuppressive agents for treatment within 3 months before screening;
6. Those whose ALT, AST or total bilirubin content goes beyond 1.5 times above normal upper limit;
7. Those who suffer from combined critical complications such as serious infection or other severe organ disease or dysfunction;
8. Pregnant or lactating women;
9. Those who are known to be allergic to drugs under trial or relevant products;
10. Those who participated in other clinical trials within 3 months before inclusion;
11. The patients who cannot comply with the research proposal as determined by the supervising physician.

Exit criteria

1. Those with incomplete or partial relieved proteinuria for 6 months after treatment;
2. Patients or their legal guardians voluntarily requests to withdraw;
3. Those against the inclusion criteria and exclusion criteria;
4. Those who need to take medications prohibited by the trail;
5. Those with poor compliance or stopping the drug for over 2 weeks;
6. Those with uncontrollable infection;
7. Those whit elevated blood glucose during the treatment, which is still difficult to control after routine treatment by endocrinologists;
8. In the TAC group, the eGFR decreased by >30%, the TAC dose was halved. And the drug concentration and renal function were reviewed after 2 weeks. If the eGFR decreased by <30%, it will continue to be used; if the eGFR still decreased by >30%, the TAC dose continues to halve, or give a minimum dose of 0.5mg / d. And the drug concentration and renal function were reviewed after 2 weeks. If the eGFR decreased by <30%, TAC will continue to be used, otherwise stop the drug;
9. Those whose ALT, AST or bilirubin rises to more than 2 times the upper limit of normal value after treatment, and continues to increase for 2 weeks; those whose ALT, AST or bilirubin rises to more than 2 times the upper limit of normal value after 2 weeks of treatment with liver protection, the drug will be discontinued. If it cannot be recovered after 2 weeks, the patient will withdraw;
10. Those with other unexplained severe comorbidities;
11. Those with pregnancy during treatment;
12. For security reasons, the research sponsor proposed to stop the study;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2018-11-26 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate of 24-hour urine protein | At week 48
  The proportion of patients with complete remission of 24-hour urine protein in the total evaluated patients. Evaluation criteria of complete remission: post-therapy urine protein level is <0.3g/24h.

SECONDARY OUTCOMES:
Partial remission remission rate of 24-hour urine protein | At week 48
  The proportion of patients with partial remission of 24-hour urine protein in the total evaluated patients. Evaluation criteria of partial remission: post-therapy urine protein decline is >50% compared with the peak value.
PLA2R antibody negative conversion rate | At week 48
  The proportion of patients with PLA2R antibody negative conversion in the total evaluated patients. Evaluation criteria of negative conversion: PLA2R antibody level is <20RU/ml.
Number of patients with adverse events | Up to 48 weeks
  Number of patients with adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xinhua Hospital affliated to Shanghai Jiao Tong University, School of Medicine, Shanghai, China